CLINICAL TRIAL: NCT00894452
Title: Factors Associated With the Variance of Oral Methadone Dosage at Steady State of Maintenance Treatment: Description of Bio-markers of Phenotype and Genotype.
Brief Title: Variance of Oral Methadone Dosage: Description of Implicated Factors
Acronym: METHADOSE
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P070603
Record Dates: First submitted 2009-03-31; First posted 2009-05-07 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Heroin Dependence
Keywords: Methadone; CYP; OPRM1; MDR1; COMT; Midazolam challenge
MeSH Terms: conditions — Heroin Dependence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — serum: orosomucoid, methadone dosage, OH midazolam/midazola ratio
  DNA: CYPs, MDR1, OPRM1, COMT
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to describe clinical, pharmacokinetic and genetic factors associated with the variance of oral methadone dosage for patients at the steady state of heroin dependence maintenance treatment. The hypothesis is that the investigators can predict 70% of the variance with few factors, including CYP 3A4 function measured with oral midazolam challenge.

DETAILED DESCRIPTION:
Patients at the steady state of methadone maintenance treatment may receive oral dosage ranging from 5 to 130 mg per day in our clinical practice. This study is aimed at providing a comprehensive cross-sectional description of factors involved in this variance:

* comorbidity with addictive and psychiatric disorders
* severity of pre-existing heroin dependence
* function of CYP 3A4 enzyme assessed with oral midazolam challenge
* genetic polymorphisms of enzymes implicated in methadone pharmacokinetic and pharmacodynamic (CYPs, MDR1, OPRM1, COMT)

The expected result is a predictive equation of oral methadone dosage at steady state.

ELIGIBILITY:
Inclusion Criteria:

* heroin dependence
* under maintenance treatment with methadone
* at steady state: stable oral methadone dosage since 3 months at least

Exclusion Criteria:

* current heroin dependence or abuse
* current cocaine and/or alcohol and/or sedatives dependence
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Defined population: participants or population are selected based on predefined criteria
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2008-12; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Functional activity CYP3A4 | Day15
  Functional activity CYP3A4 as measured by the ratio of metabolite / parent drug provided by the functional test the oral midazolam.

CONTACTS AND LOCATIONS:
Overall Officials: Florence VORSPAN, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- hospital Lariboisière-Fernand-WidalCity: PARIS, Paris, France

REFERENCES:
- [Result] Hajj A, Ksouda K, Peoc'h K, Curis E, Messali A, Deveaux LL, Bloch V, Prince N, Mouly S, Scherrmann JM, Lepine JP, Laplanche JL, Drici MD, Vorspan F. KCNH2 polymorphism and methadone dosage interact to enhance QT duration. Drug Alcohol Depend. 2014 Aug 1;141:34-8. doi: 10.1016/j.drugalcdep.2014.04.027. Epub 2014 May 14. PMID 24875677
- [Result] Icick R, Peoc'h K, Ksouda K, Bloch V, Laplanche JL, Lepine JP, Bellivier F, Vorspan F. OPRM1 polymorphism and lifetime suicide attempts among stabilized, methadone-maintained outpatients. Psychiatry Res. 2014 Aug 15;218(1-2):259-60. doi: 10.1016/j.psychres.2014.04.035. Epub 2014 Apr 24. No abstract available. PMID 24813900
- [Result] Mouly S, Bloch V, Peoc'h K, Houze P, Labat L, Ksouda K, Simoneau G, Decleves X, Bergmann JF, Scherrmann JM, Laplanche JL, Lepine JP, Vorspan F. Methadone dose in heroin-dependent patients: role of clinical factors, comedications, genetic polymorphisms and enzyme activity. Br J Clin Pharmacol. 2015 Jun;79(6):967-77. doi: 10.1111/bcp.12576. PMID 25556837
- [Result] Karsinti E, Fortias M, Dupuy G, Ksouda K, Laqueille X, Simonpoli AM, Touzeau D, Avril E, Orizet C, Belforte B, Coeuru P, Polomeni P, Icick R, Jarroir M, Bloch V, Scott J, Lepine JP, Bellivier F, Vorspan F. Anxiety disorders are associated with early onset of heroin use and rapid transition to dependence in methadone maintained patients. Psychiatry Res. 2016 Nov 30;245:423-426. doi: 10.1016/j.psychres.2016.04.064. Epub 2016 Jul 19. PMID 27620325
- [Result] Marie-Claire C, Crettol S, Cagnard N, Bloch V, Mouly S, Laplanche JL, Bellivier F, Lepine JP, Eap C, Vorspan F. Variability of response to methadone: genome-wide DNA methylation analysis in two independent cohorts. Epigenomics. 2016 Feb;8(2):181-95. doi: 10.2217/epi.15.110. Epub 2016 Jan 21. PMID 26792095
- [Result] Icick R, Peoc'h K, Karsinti E, Ksouda K, Hajj A, Bloch V, Prince N, Mouly S, Bellivier F, Lepine JP, Laplanche JL, Vorspan F. A cannabinoid receptor 1 polymorphism is protective against major depressive disorder in methadone-maintained outpatients. Am J Addict. 2015 Oct;24(7):613-20. doi: 10.1111/ajad.12273. Epub 2015 Sep 1. PMID 26331953
- [Derived] Icick R, Vorspan F, Karsinti E, Ksouda K, Lepine JP, Brousse G, Mouly S, Bellivier F, Bloch V. Gender-specific study of recurrent suicide attempts in outpatients with multiple substance use disorders. J Affect Disord. 2018 Dec 1;241:546-553. doi: 10.1016/j.jad.2018.08.076. Epub 2018 Aug 13. PMID 30153638